CLINICAL TRIAL: NCT05497440
Title: Clinical Evaluation of the All'InCath Contrast Balloon Catheter 035M When Used for Peripheral Vasculature Percutaneous Transluminal Angioplasty.
Brief Title: Evaluation of All'InCath in Peripheral Vasculature Percutaneous Transluminal Angioplasty.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough product.
Sponsor: NexStep Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-0003
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All'InCath CBC 035M Balloon Dilatation Catheter (Experimental): All participants will undergo the same intervention. Peripheral Vasculature Percutaneous Transluminal Angioplasty and Control Angiography.
  Interventions: Device: All'InCath CBC 035M Balloon Dilatation Catheter

INTERVENTIONS:
Device: All'InCath CBC 035M Balloon Dilatation Catheter — All participants will undergo the same intervention. Peripheral Vasculature Percutaneous Transluminal Angioplasty and Control Angiography.

SUMMARY:
The objective of this post-market clinical study is to obtain additional data on the safety and performance of the All'InCath 035M Balloon Dilatation Catheter when used per its Instructions for Use (IFU) during percutaneous transluminal angioplasty procedures in clinical practice.

DETAILED DESCRIPTION:
The All'InCath Contrast Balloon Catheter 035M Balloon Dilatation Catheter has received 510(k) clearance for Percutaneous Transluminal Angioplasty in the peripheral vasculature, for the treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistulae, and angiographic visualization of the vasculature when combined with the delivery of radiopaque contrast media (K191275).

The objective of this post-market clinical study is to obtain additional data on the safety and performance of the All'InCath 035M Balloon Dilatation Catheter, including device-related perioperative adverse events, vascular patency, visualization of the target area, duration of intervention, level of radiation exposure, dose of contrast agent, post-procedural adverse events and physician's feedback, when used per its Instructions for Use (IFU) during percutaneous transluminal angioplasty procedures in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be eligible to participate in the study if all of the following apply:
* Ability to provide Informed Consent

  * Can also be executed by the legal designated representative or the witness
* As per the Principal Investigator's practices as per standard of care, the subject is indicated for PTA in the peripheral vasculature, including iliac, femoral, popliteal, and renal arteries, and any treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistulae.
* Male or female >18 years old.
* Life expectancy >1 year

Exclusion criteria

The following subjects will be excluded from the study if any of the following criteria are met:

* Unstable coronary artery disease or any other uncontrolled comorbidity.
* Myocardial infarction or stroke within two (2) months before baseline evaluation.
* Previous peripheral bypass or procedure that includes the target vessel.
* Known, untreated allergy or other contraindications to contrast agents or medications used during or after PTA.
* Non-correctable bleeding diathesis, platelet dysfunction, thrombocytopenia, or any other known coagulopathy.
* The use of antiplatelet or anticoagulant therapy is contraindicated.
* Any planned major surgical or interventional procedure within 30 days after the study procedure.
* Females who are breast-feeding or child-bearing potential and not using a medically reliable method of contraception (as defined below) for the entire study duration:

  * medically reliable contraception defined as: oral, injectable, or implantable contraceptives, intrauterine contraceptive devices, or those not using another method deemed by the Investigator to be sufficiently reliable.
  * subjects who are surgically sterilized / hysterectomized or post-menopausal for longer than two (2) years are not considered childbearing potential.
* Positive pregnancy test result in women of child bearing potential or is breast-feeding.
* Incapacitated individuals and those with psychiatric disorders that could interfere with the provision of informed consent, completion of tests, therapy, follow-up or general study compliance.
* Participation in another study with investigational drug or device within the 30 days preceding and during the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Periprocedural Serious adverse events | During procedure
  Freedom from device related periprocedural adverse events and complications during PTA procedure (e.g., loss of guidewire, misdirection of catheter, vessel wall perforation or dissection requiring treatment).
Vascular patency | immediately post-procedure
  Vascular patency immediately post-procedure with adequate capability to ensure injection medium contrast into the vessel with a good visualization of the targeted area.

SECONDARY OUTCOMES:
Duration of the intervention (PTA) | Time of the procedure
  Performance of the All'InCath Contrast Balloon Catheter 035M
Level of radiation exposure during PTA (mGy). | During procedure
  Efficiency and Safety of the All'InCath Contrast Balloon Catheter 035M
Dose of contrast agent injected at the targeted location (mL). | During procedure
  Safety and performance of the All'InCath Contrast Balloon Catheter 035M
Investigator's feedback | During procedure
  Evaluation of the function of the All'InCath Contrast Balloon Catheter 035M
Major adverse events during hospitalization until discharge | before hospital discharge or 24hours after the index-procedure which ever occurs first
  Safety of the All'InCath Contrast Balloon Catheter 035M

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Chaer, Principal Investigator — UPMC 200 Lothrop Street Pittsburgh, PA 15213
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Information about subjects will be considered confidential. Subject's identification must be anonymized at the site by the Investigator or designee, when completing the case report form (CRF), study-related worksheets, preparation of clinical reports or the preparation of subject medical records. Only authorized personnel might have access to these confidential files. Every reasonable effort will be made to protect the confidentiality of the subjects throughout the study.